CLINICAL TRIAL: NCT04207229
Title: Post-Market Clinical Follow-up Registry of Patients With CODMAN CERTAS Plus Programmable Valves
Brief Title: CERTAS Programmable Valve Registry
Acronym: CERTAS
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Other Study IDs: C-CERTAS-001
Record Dates: First submitted 2019-11-27; First posted 2019-12-20 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Hydrocephalus; NPH (Normal Pressure Hydrocephalus); IIH - Idiopathic Intracranial Hypertension
MeSH Terms: conditions — Hydrocephalus; Hydrocephalus, Normal Pressure; Pseudotumor Cerebri

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- CODMAN CERTAS Programmable Valves: CODMAN CERTAS Plus Programmable Valve, CODMAN CERTAS Plus Small Inline Programmable Valve, and CODMAN CERTAS Plus Right Angle Programmable Valve.
  Interventions: Device: CODMAN CERTAS Programmable Valves

INTERVENTIONS:
Device: CODMAN CERTAS Programmable Valves — Patients will undergo implantation of the CODMAN CERTAS Plus Programmable Valve according to the device label.

SUMMARY:
Post-Market Clinical Follow-up Registry of Patients with CODMAN CERTAS Plus Programmable Valves.

DETAILED DESCRIPTION:
The CODMAN CERTAS Plus Programmable Valve is a single use implantable device designed for shunting cerebrospinal fluid (CSF) for the treatment of hydrocephalus.

The clinical investigation specifically aims to collect data on the performance measures outlined below. Data will be collected per standard of care, given the nature of the clinical investigation to capture real world data (registry); timing, frequency, and methodology of assessing the performance outcomes may therefore differ per center, subject, and/or visit.

1) Improvement of the following symptoms related to hydrocephalus:

* Gait disturbances;
* Spatial impairment;
* Cognitive abilities;
* Urinary incontinence;
* Pain caused by headaches;
* Visual acuity.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18-80 years old at time of enrollment) undergoing implantation of the CODMAN CERTAS Plus Programmable Valve according to the device label.
2. Patients willing and able to understand and sign informed consent.

Exclusion Criteria:

N/A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will receive the CODMAN CERTAS Plus Programmable Valve type most applicable for their condition, as determined by their clinician.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Performance Endpoints | 1 month, 3 months, 6 months, 12 months, 24 months, and 36 months
  The change from baseline for the following symptoms related to hydrocephalus, e.g. gait disturbances, spatial impairment, cognitive abilities, urinary incontinence, pain caused by headaches and visual acuity.

SECONDARY OUTCOMES:
Device Deficiencies | 1 month, 3 months, 6 months, 12 months, 24 months, and 36 months
  Incidence and nature of device deficiencies

OTHER OUTCOMES:
Safety Endpoints: Incidence and nature of adverse device effects | 1 month, 3 months, 6 months, 12 months, 24 months, and 36 months
  Incidence and nature of adverse device effects

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Ilic, MD, Study Director — Integra LifeSciences
Locations (8):
- Germany (7):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - UniversitätsKlinikum Essen, Essen
  - Freiburg University Hospital, Freiburg im Breisgau
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum rechts der Isar Technischen Universitat München, München
  - München Klinik Bogenhausen, München
  - Klinikum der LandesHauptStadt Stuttgart gKAôR, Stuttgart
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No